CLINICAL TRIAL: NCT00894621
Title: Norepinephrine as Early Vasopressor Therapy in Children Undergoing Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unidade de Terapia Intensiva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Noradrenalina precoce em UTIP
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Shock; Mechanical Ventilation
Keywords: Shock; Respiration, artificial; Norepinephrine
MeSH Terms: conditions — Shock; Respiratory Aspiration | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Norepinephrine (Experimental)
  Interventions: Drug: Norepinephrine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norepinephrine — Solution administration contend titrated norepinephrine in doses of 0,1 to 0,4 mc/kg/min. Initiated solution 24 hours after beginning mechanical ventilation. Use of the solution during 72 hours.
  Arms: Norepinephrine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness from early infusion of norepinephrine in pediatric patients submitted to mechanical ventilation for the use of sedative and analgesics drugs.

ELIGIBILITY:
Inclusion Criteria:

* Children, who, in the arrival or during the admission in pediatric intensive care unit, develop the need for mechanical ventilation and continuous infusion of sedatives and/or analgesics

Exclusion Criteria:

* Patients after cardiac arrest
* Patients with tracheostomy
* Patients with renal and/or hepatic failure
* Patients with previous episode of cardiac arrythmia
* Patients with mechanical ventilation forecast lesser that four days

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-11

PRIMARY OUTCOMES:
To compare norepinephrine and placebo as initial therapy in pediatric patients submitted to the mechanical ventilation with reference to hemodynamic parameters, diuresis and diuretics' use. | 5 days

SECONDARY OUTCOMES:
To assess possible side effects related with the early norepinephrine infusion. | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Geral, Caxias do Sul, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Piva J, Alquati T, Garcia PC, Fiori H, Einloft P, Bruno F. Norepinephrine infusion increases urine output in children under sedative and analgesic infusion. Rev Assoc Med Bras (1992). 2014 May-Jun;60(3):208-15. doi: 10.1590/1806-9282.60.03.008. PMID 25004265